CLINICAL TRIAL: NCT07047196
Title: A Randomized, Single-Blind, Active-controlled, Multicenter Clinical Study Evaluating the Efficacy and Safety of Intra-articular Injection of HS-20116 in Patients With Knee Osteoarthritis
Brief Title: Evaluating the Efficacy and Safety of Intra-articular Injection of HS-20116 in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-20116-301
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis,Hansoh, Chitosan Solution for Intra-Articular Use
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20116 (Experimental): HS-20116 administered as a single intra-articular injection (3 mL per dose)
  Interventions: Device: HS-20116
- Medical Chitosan (for intra-articular injection) (Active Comparator): Medical Chitosan administered as 2-3 intra-articular injections (2-3 mL per dose) in total.
  Interventions: Device: Medical Chitosan (for intra-articular injection)

INTERVENTIONS:
Device: HS-20116 — Innovative chitosan-based biomaterial intended for intra-articular injection
  Arms: HS-20116
Device: Medical Chitosan (for intra-articular injection) — Medical chitosan for intra-articular injection
  Arms: Medical Chitosan (for intra-articular injection)

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of HS-20116 for intra-articular use in patients with symptomatic knee osteoarthritis.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, active-controlled, multicenter clinical study to evaluate the efficacy and safety of intra-articular injection of HS-20116 in patients with knee osteoarthritis. Eligible subjects after screening will be randomized in a 1:1 ratio into the test group and the control group. Test group subjects will receive a single intra-articular injection of HS-20116 (3 mL) into the treated knee on Day 0. Control group subjects will receive 2-3 intra-articular injections of chitosan (2-3 mL each) on Day 0 and Day 14, with an optional injection on Day 28. The primary endpoint is the change from baseline in WOMAC pain score at Week 12 after the first injection. Each subject may choose to participate in an optional long-term follow-up visit between Weeks 22 and 28.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 40-85 years (inclusive);
2. Body mass index (BMI) ≤ 35 kg/m2;
3. Primary knee osteoarthritis in accordance with the clinical and radiological diagnostic criteria of the American College of Rheumatology (ACR), unilateral or bilateral femorotibial arthritis, with or without patellofemoral arthritis;
4. A radiographic Kellgren and Lawrence (K&L) grade of II to III in the treated knee within 6 months prior to randomization;
5. Recurrent knee pain for at least 6 months at screening, with no or poor response to the first-line oral non-opioid analgesics and non-steroidal anti-inflammatory drugs (NSAIDS);
6. After a washout period of 48 h for analgesics, the degree of pain before bilateral knee injection was assessed using the WOMAC pain score (5-grade Likert method) prior to randomization, which should meet the following criteria:

   * Treated knee: WOMAC pain score of 7-17, of which item A1 was at least 2;
   * Non-treated knee: WOMAC pain score of no more than 6.
7. Completely free to move;
8. Willing to undergo a 48-h analgesic washout period prior to visit;

Exclusion Criteria:

1. Concomitant synovial chondromatosis and villonodular synovitis of the knee;
2. Patellofemoral osteoarthritis only, where symptoms including pain mostly originated from the patellofemoral joint (patellofemoral pain syndrome);
3. Onset of clinically significant knee effusion, knee inflammation or associated symptoms, or abnormal gross examination or volume of synovial fluid at the time of joint aspiration on the day of injection;
4. Obvious varus or valgus deformity of the treated knee after clinical evaluation or imaging evaluation as judged by the investigator;
5. Concomitant autoimmune diseases, autoinflammatory diseases, or infectious arthritis, such as rheumatoid arthritis, psoriatic arthritis, articular chondrocalcinosis, gout, ankylosing spondylitis, and lupus erythematosus;
6. Other concomitant pathological changes affecting joint treatment/evaluation, such as arthrodysplasia, ipsilateral hip osteoarthritis, aseptic bone necrosis, acromegaly, Paget's disease, hemophilia, hemochromatosis, lumbosacral radicular pain, femoral nerve or sciatic nerve radicular pain, venous or lymphatic obstruction, arteritis, tendon disorder, etc.;
7. Skin infection, skin lesions, or chronic dermatosis at the puncture site;
8. Any knee injury, surgical history, or arthroscopy and treatment within 6 months prior to screening; or any surgery or other invasive operation expected to be performed during the trial;
9. Prior injection with hyaluronic acid into the treated knee within 6 months prior to randomization.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score | 12 weeks after the first injection.
  Change from baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score at Week 12 after the first injection.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Fan, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated hospital of nantong university, Nantong, China

IPD SHARING:
Plan to Share IPD: No